CLINICAL TRIAL: NCT06617234
Title: A Comparative Pilot Study on the Effectiveness of Cardiac Rehabilitation Referral Guided by Nurse-Led and LINE Robot Interventions
Brief Title: A Comparative Pilot Study on the Effectiveness of Nurse-Led and LINE Robot-Guided Cardiac Rehabilitation Referrals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202407179RINB
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Rehab; Referral; LINE Robot Intervention
Keywords: cardiac rehabilitation; automated system or chatbot

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nurse-led Intervention Program (Experimental): This intervention consists of a face-to-face educational session led by a nurse, focusing on the importance of cardiac rehabilitation. The session lasts 15-20 minutes and is tailored to the patient's medical condition and lifestyle, with follow-up reminders and personalized guidance for rehabilitation participation.
  Interventions: Other: Nurse-led Intervention Program
- LINEbot Automated Robot System (Experimental): This intervention uses the LINEbot system to send automated push notifications to participants, including educational messages, reminders for cardiac rehabilitation appointments, and health tracking prompts. Participants can log their daily health data through the system, which offers personalized advice on diet, exercise, and medication management.
  Interventions: Other: LINEbot Automated Robot System
- Control Group (Usual Care) (No Intervention): Participants in this group will receive usual care. This includes clinical evaluations by cardiologists and standard rehabilitation referrals without any specialized education or reminders. Their participation in cardiac rehabilitation will not be monitored or actively encouraged beyond routine clinical care. The patients decide independently whether or not to attend cardiac rehabilitation sessions.

INTERVENTIONS:
Other: Nurse-led Intervention Program — Nurse-led Intervention Program: This intervention consists of a face-to-face educational session led by a nurse, focusing on the importance of cardiac rehabilitation. The session lasts 15-20 minutes and is tailored to the patient's medical condition and lifestyle, with follow-up reminders and personalized guidance for rehabilitation participation.
  LINEbot Automated Robot System: This intervention uses the LINEbot system to send automated push notifications to participants, including educational messages, reminders for cardiac rehabilitation appointments, and health tracking prompts. Participants can log their daily health data through the system, which offers personalized advice on diet, exercise, and medication management.
  Arms: Nurse-led Intervention Program
Other: LINEbot Automated Robot System — Participants in this group will use the "LINEbot" automated robot system, which sends push notifications through the LINE app. The system delivers education messages, exercise guidance, and health tracking prompts. It provides daily reminders for cardiac rehabilitation participation, as well as customized messages on health management, such as diet, medication, and self-care. The system also allows users to log health data like blood pressure and heart rate.
  Arms: LINEbot Automated Robot System

SUMMARY:
The goal of this pragmatic randomized trial is to compare the effectiveness of nurse-led versus LINE bot-guided strategies on patient referrals for cardiac rehabilitation in patients with acute myocardial infarction, heart failure, or status post coronary artery bypass surgery, aged 18 years and older. The main questions it aims to answer are:

Does a nurse-led referral strategy increase cardiac rehabilitation referrals, attendance, and participation compared to routine care? Can a LINE bot-guided system improve cardiac rehabilitation referrals, attendance, and participation? Researchers will compare Intervention Group A (nurse-led face-to-face education), Intervention Group B (LINE bot automated referral system), and a Control Group (routine care) to see if nurse-led or LINE bot strategies are more effective in increasing referrals, attendance, and participation in cardiac rehabilitation programs.

Participants will:

Be randomly assigned to one of three groups. Participate in either nurse-led education, receive automated LINE bot reminders, or undergo standard care.

Have their cardiac rehabilitation referrals, attendance, and participation tracked for 12 weeks post-discharge through the hospital's medical record system.

This study seeks to provide healthcare professionals with evidence-based strategies for improving cardiac rehabilitation processes and enhancing patient engagement in rehabilitation programs.

DETAILED DESCRIPTION:
This comparative pilot study aims to evaluate the effectiveness of cardiac rehabilitation (CR) referral systems using two different intervention strategies: nurse-led education and LINE robot-guided interventions. The study's objective is to assess whether these methods can improve referral rates, attendance, and participation in CR programs compared to standard care.

Background:

Cardiovascular diseases (CVD) account for a significant proportion of global deaths and have remained the second leading cause of death in Taiwan for many years. Despite the proven benefits of CR-such as reducing mortality rates by 13%-24%, improving physical activity, enhancing cardiac function, and lowering healthcare costs-its implementation is far from ideal. International data suggest that only 20%-25% of eligible patients actually participate in CR programs.

CR is recommended for a wide range of cardiac conditions, including acute myocardial infarction (AMI), coronary artery bypass grafting (CABG), and heart failure (HF). Effective referral mechanisms are critical for ensuring that patients have access to these services. However, referral rates for CR are significantly lower than other secondary prevention measures, such as medication adherence.

Study Design and Interventions:

The study adopts an open-label, three-arm, parallel-group randomized controlled design. Participants will be randomly assigned into one of three groups:

Intervention Group A: Nurse-led education and referral program. Intervention Group B: LINE robot-guided referral system. Control Group: Standard care (usual care with CR referral as per existing practice).

Nurse-Led Education Program (Group A): Patients will receive a face-to-face education session with a trained nurse, specializing in cardiology, on the third day post-admission or after being transferred to a general ward. This session will last for 15-20 minutes and will cover the following key areas:

The importance of CR in improving cardiac function, reducing rehospitalization rates, and enhancing quality of life.

The structure of hospital-based CR programs and how they combine exercise monitoring, diet management, emotional support, and medication management.

Individualized discussions, where patients can ask questions and receive tailored advice based on their medical history and lifestyle.

LINE Robot-Guided Program (Group B): This intervention uses the LINEbot system, designed to automate patient education and reminders. The system sends daily messages to patients, including CR-related educational content, exercise instructions, and motivational prompts. Features include:

Automated educational messages: covering CR importance, exercise guidance, and diet management.

Exercise tracking: allowing patients to log their physical activities and vital signs.

Communication tools: enabling interaction between patients and the healthcare team.

Study Duration and Data Collection: The study will last 12 weeks for each participant. Data will be collected from hospital records, patient self-reports, and the automated LINE system. Outcomes measured will include:

Primary Outcomes: Referral rates, attendance at CR sessions, and program completion.

Secondary Outcomes: Patient satisfaction, perceived usefulness of the intervention, and health improvements (e.g., physical activity, heart rate variability).

Randomization and Recruitment: Participants will be recruited from cardiology wards based on inclusion criteria (patients diagnosed with AMI, HF, or post-CABG with NYHA Class I-III). Randomization will be performed using the REDCap system, with stratification by diagnosis (AMI, HF, or post-CABG).

Significance: This study will provide critical insights into the effectiveness of nurse-led and digital interventions in increasing participation in CR programs. It will explore the potential of digital tools like LINEbot in enhancing patient engagement, potentially reducing the workload of healthcare providers while promoting patient self-management and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≧18 years old
* AMI(STEMI or NSTEMI after PCI)
* Heart failure with New York Heart Association (NYHA) functional class I-III .
* After coronary artery bypass surgery (CABG)
* Patients must have a smartphone with internet
* Able to use the LINE messaging (send and receive messages)

Exclusion Criteria:

* Cardiac rehabilitation absolute or relative contraindications.
* Acute decompensated heart failure, New York Heart Association (NYHA) functional class IV
* Cognitive impaired
* Without smartphones
* Attending physician finds it unsuitable.
* One patient was enrolled in the same ward

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-01-30 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Cardiac Rehabilitation Participation Rate | 12 weeks post-discharge
  The percentage of patients who are referred to and actively engage in cardiac rehabilitation programs after discharge. Active participation is defined as attending at least one session of a cardiac rehabilitation program within the 12-week period following discharge from the hospital.

IPD SHARING:
Plan to Share IPD: No
At this time, there is no plan to share individual participant data (IPD) due to concerns about maintaining participant privacy and confidentiality. The study involves sensitive health information, and ensuring the protection of participant identity is a priority.

REFERENCES:
- [Result] Clark AM, King-Shier KM, Duncan A, Spaling M, Stone JA, Jaglal S, Angus J. Factors influencing referral to cardiac rehabilitation and secondary prevention programs: a systematic review. Eur J Prev Cardiol. 2013 Aug;20(4):692-700. doi: 10.1177/2047487312447846. PMID 23847263